CLINICAL TRIAL: NCT03430869
Title: Exploring and Subtyping the Pathophysiology of Neurodegeneration in Late-life Depression: Implications for Treatment and Prognosis in the Future
Brief Title: Pathophysiology of Neurodegeneration in Late-life Depression (AV45+THK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201601655A0
Record Dates: First submitted 2017-11-20; First posted 2018-02-13 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder
Keywords: late-life depression; major depressive disorder; Alzheimer's disease dementia; neurodegeneration; amyloid plague, tau protein
MeSH Terms: conditions — Depressive Disorder, Major; Nerve Degeneration; Frontotemporal Dementia | interventions — florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F-18 AV-45 (Experimental): F-18 AV-45 imaging
  Interventions: Drug: F-18 AV-45
- F-18-THK-5351 (Experimental): F-18-THK-5351 imaging
  Interventions: Drug: F-18-THK-5351

INTERVENTIONS:
Drug: F-18 AV-45 — In the present project, the investigators will recruit 40 patients with lifetime major depressive disorder, and 20 non-depressed cognitively normal comparison subjects. Alzheimer's disease pathology (A) was determined by measuring Aβ deposition by F-18 AV-45 PET.
  Arms: F-18 AV-45
Drug: F-18-THK-5351 — In the present project, the investigators will recruit 40 patients with lifetime major depressive disorder, and 20 non-depressed cognitively normal comparison subjects. All subjects will further undergo F-18-THK-5351 image study to detect underlying tau pathology. By doing this, the investigators will elucidate the neurodegenerative pathophysiology behind the link between depressive disorder and the subsequent development of dementia.
  Arms: F-18-THK-5351

SUMMARY:
Late-life depression has been frequently associated with cognitive impairment. Several meta-analyses consistently suggested that a history of depression approximately doubles an individual's risk for developing dementia later in life. Neurodegeneration may play an important component in late-life depression. The pathophysiology behind the link between late-life depression and the subsequent development of dementia largely remains unclear, and should be heterogeneous. This highlights the need to identify specific neurodegenerative pathways involved in late-life depression, which will facilitate research on mechanisms and new treatments in the future.

The recently published the National Institute on Aging and the Alzheimer Association (NIA-AA) criteria might provide new insights and frameworks to explore the patterns of neurodegenerative process in elderly depressed patients and to categorize them into different biomarker-based groups. In the present project, the investigators will recruit 40 patients with lifetime major depressive disorder, and 20 non-depressed cognitively normal comparison subjects. Alzheimer's disease pathology (A) was determined by measuring Aβ deposition by F-18 AV-45 PET, and neurodegeneration (N) was established by measuring hippocampal volume using MRI. Individuals were categorised as A-N-, A+N-, A+N+, or suspected non-Alzheimer's disease pathophysiology (A-N+, SNAP). All subjects will further undergo F-18-THK-5351 image study to detect underlying tau pathology. By doing this, the investigators will elucidate the neurodegenerative pathophysiology behind the link between depressive disorder and the subsequent development of dementia.

DETAILED DESCRIPTION:
Visit 1, Screening assessments (Day 1)

The purpose is to determine eligibility for the proposed study. Screening period may take place over several days to one week after the first visit. Screening assessments will include:

1. Study explanations and obtainment of informed consent;
2. Inclusion and exclusion Criteria;
3. Demographics, medical history, and concomitant medications;
4. Clinical characteristic of MDD;
5. Safety measurements include vital sign, ECGs and laboratory tests. In addition, a pregnancy test will be performed at screening for females who are of childbearing potential (not for subjects with postmenopause period). A resting ECG and laboratory tests will be taken during the period of the study visit or had been done within 3 months before study visit.
6. Fertile females must avoid becoming pregnant 30 days after administration of F-18 AV-45 and 18F-THK-5351.The investigators will advise fertile females to use adequate contraceptive methods during this period, e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidal foam/gel/film/cream or occlusive cap(diaphragm or cervical/vault caps) with spermicidal foam /gel /film /cream. In addition, a pregnancy test will be performed at screening for females who are of childbearing potential (the test must be negative).This test is not applicable for female subjects with postmenopausal period; permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy.
7. Cognitive function assessment includes MMSE, CDR and comprehensive neurocognitive battery.

Visit 2, Image study (Month 1±14 days) F-18 AV-45 PET study will be conducted for all subjects. PET data will be acquired using SIMENS PET/CT or PET/MRI scanner. For PET/CT protocol, a dynamic brain PET scan will be started simultaneously with the injection of F-18 AV-45 PET after a low-dose CT scan for patient positioning and attenuation correction. Instead of PET/CT, the investigators will also consider PET/MRI for better soft tissue contrast and limited radiation exposure for multiple scan session. However, the attenuation map delineated from MRI is not consistent, and the delicate PET/MRI protocol is still under evaluation. Vital sign will be checked before and at the end of the image study for all subjects. Subjects will be continuously observed for signs of adverse events or serious adverse events. Each study participant (or their caregiver if applicable) will be contacted by phone approximately 7-14 days after the PET imaging study or at the next follow-up visit of outpatient department to confirm their well-being and query them about any new adverse events. Study-emergent AEs will be monitored till resolution or relatively stable state.

Visit 3, Image study (Month 1±14 days) All participants will receive F-18-THK-5351 PET image study. PET data will be acquired using SIMENS PET/CT or PET/MRI scanner. For PET/CT protocol, a dynamic brain PET scan will be started simultaneously with the injection of F-18-THK-5351 after a low-dose CT scan for patient positioning and attenuation correction. Instead of PET/CT, the investigators will also consider PET/MRI for better soft tissue contrast and limited radiation exposure for multiple scan session. However, the attenuation map delineated from MRI is not consistent, and the delicate PET/MRI protocol is still under evaluation. Vital sign will be checked before and after the image study. Safety measurements include ECG, and clinical labs will be performed at the end of the image study for all subjects. Subjects will be continuously observed for signs of adverse events or serious adverse events. Each study participant (or their caregiver if applicable) will be contacted by phone approximately 7-14 days after the PET imaging study or at the next follow-up visit of outpatient department to confirm their well-being and query them about any new adverse events. Study-emergent AEs will be monitored till resolution or relatively stable state.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled subjects will be 50 to 90 years of age. They should understand the content of consent and sign consent after the explanation of the benefits and possible side effects of this trial
2. Patients with a clinical diagnosis of major depressive disorder according to the DSM -5 criteria (APA, 2013).
3. Comparison subjects evaluated for lifetime absence of psychiatric illness by MINI interview (Sheehan et al., 1998).
4. Fertile females must avoid becoming pregnant and must use adequate contraceptive methods for 30 days after administration of study radiotracer.

Exclusion Criteria:

1. Any subject has clinically definite diagnosis of dementia before study recruitment according to the NIA-AA criteria for possible or probable clinically-defined AD dementia ( McKhann, 2011) or the DSM -5 criteria for any type of dementia (APA, 2013).
2. Any subject has clinically significant or unstable medical diseases including metabolic, renal, liver, lung or cardiovascular disorders including metabolic, renal, liver, lung or cardiovascular disorders
3. Any subject has a current or past history of clinically significant neurological insults affecting brain structure or function like completed stroke, head injury or epilepsy
4. Any subject has current alcohol or other substances abuse and/ or dependence within the recent one year, or previously prolonged history of substances abuse
5. Any females who is pregnant or lactating
6. General MRI, and/or PET exclusion criteria including subjects who are pregnant, or had received brain aneurysm surgery, or implanted pacemaker, mechanical valves or cochlear implant.
7. Any subjects with history of severe allergic or anaphylactic reactions particularly to the study medication, or any subjects who are recognized as high risk of adverse effects by principle investigator.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The standard uptake value ratio (SUVR) of 18F-florbetapir | three years
  The primary outcome is to measure the standard uptake value ratio (SUVR) of 18F-florbetapir in patients with major depressive disorder and compare the difference between patients and non-depressed subjects. 18F-florbetapir SUVRs of each volume of interest are analyzed using whole the cerebellum as the reference region.

SECONDARY OUTCOMES:
The standard uptake value ratio (SUVR) of 18F-THK-5351 | three years
  The secondary outcome is to measure the standard uptake value ratio (SUVR) of 18F-THK-5351 in patients with major depressive disorder and compare the difference between patients and non-depressed subjects. 18F-THK-5351 SUVRs of each volume of interest are analyzed using the pons as the reference region.

CONTACTS AND LOCATIONS:
Overall Officials: KUAN YI WU, Principal Investigator — Attending physician
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No